CLINICAL TRIAL: NCT05189899
Title: Pain's Treatment With Virtual Reality in Hemodialysis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The trial was not performed because logistical problems
Sponsor: Consorci Sanitari de l'Alt Penedès i Garraf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CSAPG-2
Record Dates: First submitted 2021-11-20; First posted 2022-01-13 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Chronic Pain; Chronic Kidney Diseases
MeSH Terms: conditions — Chronic Pain; Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Crossover clinica trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With virtual reality (Active Comparator): One hemodialysis session with virtual reality
  Interventions: Device: Virtual reality
- without virtual reality (No Intervention): One hemodialysis session without virtual reality

INTERVENTIONS:
Device: Virtual reality — One hemodialysis session with virtual reality and one other without it
  Arms: With virtual reality

SUMMARY:
Pain is a frequent and difficult to treat symptom in patients with advanced kidney disease undergoing hemodialysis. Pharmacokinetics and pharmacodynamics have complex pharmacokinetics and pharmacodynamics in these types of patients, so non-pharmacological therapies could be very useful. In this project the investigators propose to test whether the use of a virtual reality platform, designed by the company Psious and tested in other clinical settings, can reduce the pain that patients experience during connection to the dialysis session.

For this the investigators have designed a crossover clinical trial, which will be carried out on 107 hemodialysis patients, in which the intensity of pain (primary objective) and anxiety (secondary objective) that patients experience in the sessions in which participants are treated Using virtual reality, it will be compared with the intensity of pain and anxiety experienced by these same patients, in sessions in which the virtual reality platform is not used.

The results of this clinical trial can support the use of virtual reality as an adjunctive pain treatment in patients with advanced kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis for at least 3 months
* Pain for for at least 3 months
* Signature of informed consent

Exclusion Criteria:

* Pain from a traumatology disease
* Formal diagnose of dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-04-15 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Pain measured by using the revised Faces Pain Scale - Revised (FPS-R) | From the moment of connection to dialysis until 30 minutes later
  Pain measured by using the revised Faces Pain Scale - Revised (FPS-R). The scale ranges from 0 to 10, with 0 being the absence of pain and 10 being the maximum pain

SECONDARY OUTCOMES:
Anxiety measured by using the Hamilton scale | From 1 hour before dialysis connection to 30 minutes after
  Anxiety measured by using the Hamilton scale. The scale ranges from 0 to 56, being 56 the maximun level of anxiety.